CLINICAL TRIAL: NCT01417689
Title: Eyedrop Instillation Technique: A Randomizaed Controlled Trial
Brief Title: Eyedrop Instillation Technique
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oftalmologia Hospital Sotero del Rio (Other)
Responsible Party: Eugenio A. Maul, 1 Pontificia Universidad Catolica de Chile, 2 Hospital Sotero del Rio.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Oftalmo_Glaucoma_001
Record Dates: First submitted 2011-08-15; First posted 2011-08-16 (Estimated); Last update posted 2011-08-16 (Estimated); Status verified 2011-08

CONDITIONS: Glaucoma; Glaucoma Suspect
Keywords: glaucoma; randomized controlled trial; eye drops; instillation; compliance
MeSH Terms: conditions — Glaucoma; Ocular Hypertension; Patient Compliance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Open-eyes (Active Comparator): Patients in this arm are encourage to attempt eye drop instillation using the most commonly used technique that involves looking up, pulling inferior lid down and putting the drop in the inferior cul de sac.
  Interventions: Other: Encouragement to attempt eye drop instillation with a specific technique
- Closed-eyes (Experimental): Patients in this group are encouraged to attempt eye drop instillation with both eyes closed near the medial canthal region. After feeling contact with the drop on the skin the drop is expected to enter the eye when opening the eye and resuming blinking.
  Interventions: Other: Encouragement to attempt eye drop instillation with a specific technique

INTERVENTIONS:
Other: Encouragement to attempt eye drop instillation with a specific technique — Encouragement to one of the 2 techniques (open eyes and closed eyes) is accomplished through a standardized educational session designed to take2-5 minutes.

SUMMARY:
Eye drop instillation is a problem from glaucoma patients. Studies reveal that 30-50% of glaucoma patients have problems instilling their eyedrops. These problems include not hitting the eye, spending many drops to get a single successful instillation and bottle contamination.

The present study will evaluate the effect of encouraging patients to put their eyedrops using one of 2 techniques, randomly assigned, to determine which is more successful at instilling the eye drop into the eye while spending the least amount of drug.

In one of the techniques the patient instills the eye drop with their eyes open in the inferior cul de sac. In the other technique the patient instills the eye drop with the eyes closed near the inner canthal region.

Patients will be randomized to encouragement to use the drops with either of the techniques. Encouragement will take place over a visit where they will be subjected to:

* Baseline evaluation of eye drop instillation using their usual technique.
* Short (2-5 minute) educational session session for the assigned technique.
* Followup evaluation immediately after the educational session.

ELIGIBILITY:
Inclusion Criteria:

* Glaucoma or glaucoma suspect
* Use of topical glaucoma medication in both eyes for at least 1 year prior to enrollment
* VA of 20/60 or better with habitual correction in at least one eye

Exclusion Criteria:

* Previous history of allergy to fluorescein
* Received topical anesthesia for IOP measurement or other reason within the last 2 hours.
* Rejects participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2011-08; Primary Completion 2011-12 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Complete success | Day 1. Immediately after intervention.
  Total success is defined as: Patient manages to instill one eyedrop into de eye spending only one eye drop.
  Difference in the proportion of patients achieving successful eye drop instillation in each of the 2 groups. For the main analysis the results of the first eye (Right or left randomly determined will be used) A mixed model with both eyes in the analysis will also be presented for sensitivity analysis.

SECONDARY OUTCOMES:
Qualified success | Day 1. Same day as intervention.
  Qualified success is defined as: Patient manages to instill one eye drop into the eye regardless of the amount of drops spent.
  Difference in the proportion of patients achieving successful eye drop instillation in each of the 2 groups. For the main analysis the results of the first eye (Right or left randomly determined will be used) A mixed model with both eyes in the analysis will also be presented for sensitivity analysis.
Number of drops | Day 1.
  Number of eye drops spent on attempted instillation in the first eye (randomly assigned). The average number of drops spent on each of the groups will be compared.
  Mixed models with data from both eyes will also be presented for sensitivity analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Eugenio A Maul, MD MPH, Principal Investigator — Pontificia Universidad Catolica de Chile. Hospital Sotero del Rio.
Locations (1):
- Hospital Sotero del Rio, Santiago, RM, Chile